CLINICAL TRIAL: NCT07075081
Title: The Protective Role of Ceremony Against Substance Use for American Indian Adults
Brief Title: Gii'Igoshimong: Sitting With Your First Family
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00030209; R01DA057904 (NIH)
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Substance Use; Mental Health Issue
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: An effectiveness trial where Gii'igoshimong will be tested in a randomized waitlist control trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators, data collectors, and data analysts will be blinded to participant randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceremony (Experimental): Completes baseline, ceremony, and post assessments (in that order).
  Interventions: Other: Ceremony
- Waitlist control (No Intervention): Completes baseline, post assessments, and is offered ceremony (in that order) but is not required to complete ceremony for study involvement.

INTERVENTIONS:
Other: Ceremony — Lifecourse ceremony led by Elders that used to be offered to everyone prior to colonization
  Arms: Ceremony

SUMMARY:
The goal of this randomized wait-list control study is to understand the relationship between ceremony and substance use (SU), SU risk (e.g., SU severity, depressive symptoms) and protective factors (e.g., spirituality, community support). The main questions it aims to answer are:

* Will adults enrolled in Gii'igoshimong show improved SU outcomes compared to those in control groups?
* Will self-relevant processing networks activated during stimulus engagement increase from pre- to post- engagement in ceremony and at 6-month follow-up?

Researchers will compare adults that complete Gii'igoshimong with those that do not complete Gii'igoshimong to see if health outcomes are different.

After completing baseline assessments, participants will be randomized to complete Gii'igoshimong now (intervention) or after the participants have completed the 1 month and 6-month post assessments (waitlist control). All participants (intervention and waitlist control) within a cohort will complete 1 month and 6 month post assessments at the same time.

DETAILED DESCRIPTION:
This project seeks to engage American Indian (AI) adults with community and spiritual worldviews via ceremony (Gii'igoshimong). In doing so, the investigators will attempt to buffer the effects of historical trauma, personal trauma, and lifelong risk factors for substance use, thereby improving substance use behaviors, related outcomes, and overall health.

The Community-Based Participatory Research will enroll AI adults (Aim 2 & 3) to implement a randomized controlled trial (N = 300 target adults) with a wait-list design respectful of cultural norms of inclusion. The investigators will evaluate the relationship between ceremony and adult substance use and identify multilevel factors (i.e., psychosocial, neurocognitive) through which traditional practices convey protection against substance use. The investigators will assess and develop a menu of implementation strategies (Sub-aim 2) to support community priority of long-term sustainment of the ceremonial practice.

TRIAL (Aim 2):

An effectiveness trial where Gii'igoshimong will be tested in a randomized waitlist control trial with N = 300 participants. Once enrolled and consented into the trial, participants will complete baseline assessments. Once baseline assessments are complete, participants will be randomized into either intervention (ceremony) or control (wait-list). Intervention is an up to four-day ceremony, that was traditionally offered to every Anishinaabe person when the Anishinaabe person reached puberty. Today, this ceremony is being revived, and yet, accessibility to this ceremonial opportunity remains low. Ceremony will be described in more detail below. Both intervention and control arms will complete 1 month post and 6-month post assessments. Control arm participants will be offered the ceremony after completion of the 6-month assessments.

POST-CEREMONY FOCUS GROUP DISCUSSIONS (FGD) (Sub-aim 2) The investigators will conduct focus group discussions (FGDs) with ceremony treatment arm participants at six months post-baseline (6 total FGDs) to get participant feedback on the ceremony, thoughts on the effects of participation, and suggestions for strengthening implementation.

KEY INFORMANT INTERVIEWS (KII) (Sub-aim 2) The investigators will conduct key informant interviews (KIIs) with ceremony leaders at mid-trial to get feedback on ceremony implementation and suggestions for improving implementation moving forward.

IMPLEMENTATION MAPPING FGD (Sub-aim 2) The investigators will conduct two sequential FGDs with ceremony leaders and other community leaders. In the first implementation mapping FGD, the investigators will present the results of the KIIs/FGDs that were done during the trial, outlining what the investigators think are the key issues/barriers to implementation of the ceremony in the community moving forward. The investigators will then facilitate a group discussion where the investigators try to reach consensus on those issues. After FGD 1, the investigators will (independently) try to come up with some strategies that the tribe could use to support implementation in the long-term. In FGD 2, the investigators will present these back to the same group and get feedback/try to seek consensus

ELECTROENCEPHALOGRAPHY (EEG) (Aim 3) The investigators will examine the neurocognitive effects of Gii'igoshimong ceremony and associated stimuli relevant to reducing substance use. This study will establish the measurement validity of electroencephalography/event related potential (EEG/ERP) indicators of self-referential processing and an indicator of cultural identification, a critical step in the science of delineating the potential of cultural factors as disease modifying processes. EEG assessments will be a required activity of the Trial. These assessments will be completed at the same time as Trial survey assessments.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older
* Self-identify as Ojibwe/Anishinaabe/Chippewa
* Self-report using any kind of substances in the past 30 days
* Have no history of head injury with loss of consciousness
* Do not currently have Type 2 Diabetes
* Are not currently pregnant

Exclusion Criteria:

* 18 years of age or younger
* Does not Self-identify as Ojibwe/Anishinaabe/Chippewa
* Does not self-report using any kind of substances in the past 30 days
* Has history of head injury with loss of consciousness
* Has Type 2 Diabetes
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Days of substance use assessed by Timeline Follow Back (TLFB) | baseline, 1 month, 6 month
  Days of substance use
Flourishing Scale | baseline, 1 month, 6 month
  Score range: 8-40; lower score means higher Positive mental health
Late Positive Potential (LPP) quantified as the average EEG response in microvolts to adjectives in the Self-referential Processing Task | baseline, 1 month, 6 month
  Larger magnitude LPP (i.e., higher microvolts) indicates larger attention engagement

SECONDARY OUTCOMES:
Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | baseline, 1 month, 6 month
  Score range: 0-27; lower score is indicative of lower risk
Center for Epidemiologic Studies Depression Scale (CESDR-10) | baseline, 1 month, 6 month
  Scale range: 0-40; lower score = lower depression
General Anxiety Disorder-7 (GAD-7) | baseline, 1 month, 6 month
  Scale range: 7-28; lower scores indicates lower anxiety
Self-rated (physical, mental, spiritual) health | baseline, 1 month, 6 month
  Adapted from the Composite International Diagnostic Interview; Score ranges 1-5 for physical health; Score ranges 1-5 for mental health; Score ranges 1-5 for spiritual health; lower score is better

OTHER OUTCOMES:
Oslo Social Support Scale (OSSS) | baseline, 1 month, 6 month
  Scale range: 3-14; higher score is better
Cultural efficacy | baseline, 1 month, 6 month
  Adapted from Native Wellness Assessment; Score range: 20-28; lower score is better
Traditional Spiritual Activities score | baseline, 1 month, 6 month
  Score range: 12-24; lower score is better
Spiritual Values score | baseline, 1-month post, 6-month post
  Score range: 1-4; lower score is better

CONTACTS AND LOCATIONS:
Overall Officials: Migis Gonzalez, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Great Lakes Hub, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez MB, Johnson AZ, Martin LA, Naawakwe, Fish J, Sevillano L, Walls ML, Staples LO. Planting the seed: using research as a tool to revitalize puberty ceremonies in Anishinaabe communities. Qual Res J. 2024 Dec 4;24(5):473-490. doi: 10.1108/QRJ-03-2024-0072. Epub 2024 Oct 10. PMID 40191601